CLINICAL TRIAL: NCT06274788
Title: Title: A Single-arm, Open-label, Prospective, Multicenter Safety Study to Evaluate the Occurrence of Essential Fatty Acid Deficiency (EFAD) in Pediatric Patients With Parenteral Nutrition-associated Cholestasis (PNAC) Who Require More Than Eight Weeks of Omegaven Treatment
Brief Title: Safety Study to Evaluate the Occurrence of EFAD in Pediatric Patients With PNAC Who Require More Than Eight Weeks of Omegaven Treatment
Status: Recruiting | Type: Observational
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Other Study IDs: OMEG-054-CP4
Record Dates: First submitted 2024-01-26; First posted 2024-02-23 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-02

CONDITIONS: Parenteral Nutrition Associated Liver Disease (PNALD); Essential Fatty Acid Deficiency; Malnutrition; Pediatric ALL
MeSH Terms: conditions — Malnutrition; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — fish oil triglycerides

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single arm OMEGAVEN® (fish oil triglycerides; injectable emulsion): The dose of investigational drug (study treatment), as well as all other components of the overall nutritional regimen is solely at the discretion of the Investigator. It is assumed the Investigator will use sound medical judgement, follow institutional standards of care regarding the nutrition provided to each patient, and review applicable prescribing information indicating the maximum and recommended dose of Omegaven of 1 g/kg/day infused intravenously over 8 to 24 hours as long as the infusion rate does not exceed 1.5 mL/kg/hour.
  Interventions: Drug: Omegaven® (fish oil triglycerides) Injectable Emulsion

INTERVENTIONS:
Drug: Omegaven® (fish oil triglycerides) Injectable Emulsion — Pediatric patients Pediatric patients with new-onset PNAC
  Drug: Omegaven® (fish oil triglycerides) Injectable Emulsion Dose, frequency and duration is a decision of the Investigator

SUMMARY:
This study will demonstrate safety in pediatric patients with Parenteral Nutrition-Associated Cholestasis treated with Omegaven®, which is indicated as a source of calories and fatty acids in this patient population

ELIGIBILITY:
Inclusion Criteria:

1. Patient's parent(s) or legal guardian(s) has provided a signed and dated Informed Consent Form (ICF).
2. Pediatric patient (<18 years) has been diagnosed with PNAC, defined as direct or conjugated bilirubin (DBil) ≥ 2.0 mg/dL with no other known cause of liver dysfunction at the time of enrollment and is expected to require Omegaven treatment for at least eight weeks.
3. Patient has oral or enteral feeding intolerance or at least one gastrointestinal disorder requiring PN.

Exclusion Criteria:

1. Patient has received Omegaven within four weeks before inclusion in the study
2. Patient has any other known cause of chronic liver disease such as hepatitis C, cystic fibrosis, biliary atresia, alpha-1-antitrypsin deficiency, passive hepatic congestion due to heart failure, etc.
3. Patient has known cirrhosis (liver biopsy is not required under this protocol).
4. Patient has been previously diagnosed with, or has prior evidence of, portal vein thrombosis.
5. Patient has previously received a liver-only or liver-inclusive transplant.
6. Patient has hemodynamic instability due to any major cardiac anomaly.
7. Patient has a major life-threatening disease (e.g., sepsis requiring high-dose vasopressors, acute respiratory distress syndrome, veno-occlusive disease, cancer).
8. Patient has multi-organ failure, septic shock, hypotension requiring pressor therapy, persistent pulmonary hypertension requiring inhaled nitric oxides, or requires extracorporeal membrane oxygenation (ECMO) or similar intervention.
9. Patient has renal failure and requires renal replacement therapy.
10. Patient has a severe hemorrhagic disorder.
11. Patient has severe hyperlipidemia or a severe disorder of lipid metabolism characterized by hypertriglyceridemia (i.e., serum triglyceride level > 1,000 mg/dL).
12. Patient has a record of EFAD before inclusion in the study
13. Patient has been diagnosed with or is suspected to have an inborn error of metabolism.
14. Patient has a known hypersensitivity to fish or egg protein or to any of the active ingredients or excipients of Omegaven.
15. Patient is subject to treatment limitation.
16. Patient is enrolled in any other study with an investigational medicinal product during the course of the current study.

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Male and female pediatric patients with PNAC and expected requirement of Omegaven for at least 8 weeks will be enrolled at multiple sites; PNAC is defined as being PN-dependent with a DBil level ≥ 2.0 mg/dL and no other known cause of liver dysfunction.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of essential fatty acid deficiency (EFAD) | Up to week 56
  EFAD as defined by the triene:tetraene (T:T) ratio; severity of EFAD will be graded and analysed based on T:T ratio (suspected ≥ 0.05, moderate ≥ 0.20, and severe ≥ 0.40)

SECONDARY OUTCOMES:
Incidence of clinical EFAD | Up to week 56
  Clinical EFAD is defined by clinical symptoms (like dry, scaly rash, hair loss, hair depigmentation, poor wound healing, growth restriction, and increased susceptibility to infection) and T:T ratio ≥ 0.083
Time from treatment start to EFAD diagnosis | Up to week 56
  Time from treatment start to EFAD diagnosis
Incidence of adverse events (AEs)/serious adverse events (SAEs) | Up to week 56
  The incidence of AEs/SAEs considered by the Investigator to be related to study treatment
Routine laboratory tests: Direct or conjugated bilirubin | Up to week 56
Routine laboratory tests: triglycerides | Up to week 56
Fatty acid profiles: α-linolenic acid | Up to week 56
Fatty acid profiles: linoleic acid | Up to week 56
Fatty acid profiles: arachidonic acid | Up to week 56
Fatty acid profiles: mead acid | Up to week 56
Fatty acid profiles: oleic acid | Up to week 56
Fatty acid profiles: docosahexaenoic acid (DHA) | Up to week 56
Fatty acid profiles: eicosapentaenoic acid (EPA) | Up to week 56
Anthropometric measures: body weight | Up to week 56
Anthropometric measures: body height/length | Up to week 56
Anthropometric measures: head circumference | Up to week 56

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Memorial Health Service, Fountain Valley, California
  - University of California Los Angeles, Los Angeles, California
  - The University of Chicago, Chicago, Illinois
  - Children's Hospital Corporation d/b/a Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Board of Regents of the University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine Houston, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Seattle Children's Hospital d/b/a Seattle Children's Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No